CLINICAL TRIAL: NCT06918301
Title: Comparison of Cardiac Index and Stroke-volume-index Measured by Pulmonary Artery Catheter, FloTrac® and Argos® in Cardiac Surgery Patients.
Status: Recruiting | Type: Observational
Sponsor: Karlsburg Hospital (Other)
Responsible Party: Principal Investigator, Prof. Dr. Matthias Heringlake, Head of department of anesthesiology and intensive care, Karlsburg Hospital
Other Study IDs: KAIKB 2025-1
Record Dates: First submitted 2025-03-29; First posted 2025-04-09 (Actual); Last update posted 2025-04-09 (Actual); Status verified 2025-04

CONDITIONS: Cardiac Failure Acute; Hemodynamic Monitoring

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — blood gas analysis
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: Measurement of cardiac performance — Measurement of cardiac performance by different devices

SUMMARY:
A comparison of cardiac performance determined by stroke-volume-index measured by different mechanisms in patients during and after cardiac surgery:

1. Pulmonary artery catheter
2. Flo Trac
3. Argos Monitor Investigations will be done in theater and on ICU in ventilated and spontaneously breathing patients.

ELIGIBILITY:
Inclusion Criteria:

* Patient after cardiac surgery with pulmonary artery catheter

Exclusion Criteria:

* Hemodynamic instability, no consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients after cardiac surgery requirering a pulmonary artery catheter
Sampling Method: Non-Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2025-03-01 (Actual); Primary Completion 2025-06-01 (Estimated); Study Completion 2025-12-01 (Estimated)

PRIMARY OUTCOMES:
stroke volume index | 24 hours
  stroke volume index

CONTACTS AND LOCATIONS:
Overall Officials: Matthias Heringlake, Principal Investigator — Head of Department of Anesthesiology and intensive care, Karlsburg Hospital
Locations (1):
- Klinik für Anästhesiologie und Intensivmedizin, Klinikum Karlsburg, Karlsburg, Germany

IPD SHARING:
Plan to Share IPD: No